CLINICAL TRIAL: NCT04755751
Title: Acute and Long Term Evaluation of Exercise Capacity in Response to Enzyme Replacement Therapy in Pediatric Pompe Disease.
Brief Title: Exercise Capacity in Response to Enzyme Replacement Therapy in Pediatric Pompe Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, l_bentur, Head of Pediatric Pulmonary Institute, Rambam Health Care Campus
Other Study IDs: RMB-045-18
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Pompe Disease Infantile-Onset
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — self-collected blood samples (on a Guthrie card) for enzyme blood levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Pompe patients: A retrospective - prospective study evaluating pediatric patients with Pompe before and 2 days after ERT on multiple occasions and different dosing. Evaluation included cardiopulmonary exercise testing (CPET), 6 minute-walking test (6MWT), motor function test (GMFM-88) and self-collected blood samples (on a Guthrie card) for enzyme blood levels.
  Interventions: Diagnostic Test: Cardiopulmonary exercise testing (CPET)

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — CPET using a cycle ergometer (COSMED, Rome, Italy) beginning with a no resistance warm up lasting 1 to 3 minutes and followed with an incrementing resistance adapted to the patient's functional capacities according to the examiner's free judgment and ranging from no resistance (20 Rounds Per Minute (RPM)/minute) 5 to 20 Watts/minute on ramps or by successive stages

SUMMARY:
Our aims are to investigate the acute and long term effect of ERT on exercise capacity; comparing the effect of different ERT dosages (as prescribed by the clinician according to clinical judgment) and assessing the relationship between enzyme blood level and exercise capacity. Such evaluation may allow a more objective quantification of the response to ERT.

DETAILED DESCRIPTION:
Pompe disease is a rare autosomal recessive metabolic myopathy caused by reduced or absence activity of the lysosomal enzyme acid alpha-glucosidase (GAA). Enzyme replacement therapy (ERT) with Myozyme has significantly improved the prospect of patients with infantile Pompe disease (IPD). Most IPD patients show clinical improvement on therapy, but deteriorate at different time points, raising the possibility that increasing drug delivery might halt the progression of the disease. Data on the effects of ERT therapy on physiological variables related to exercise tolerance is scarce.

Our aims are to investigate the acute and long term effect of ERT on exercise capacity; comparing the effect of different ERT dosages (as prescribed by the clinician according to clinical judgment) and assessing the relationship between enzyme blood level and exercise capacity. Such evaluation may allow a more objective quantification of the response to ERT.

Methods: A retrospective - prospective study evaluating pediatric patients with Pompe before and 2 days after ERT on multiple occasions and different dosing. Evaluation included cardiopulmonary exercise testing (CPET), 6 minute-walking test (6MWT), motor function test (GMFM-88) and self-collected blood samples (on a Guthrie card) for enzyme blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Pompe patients >5 years that have been on alpha-glucosidase (GAA).

Exclusion Criteria:

* Oxygen saturation > 90% in room air without ventilatory assistance.
* Patients will be excluded if they required any invasive ventilation or if they required noninvasive ventilation while awake and upright

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children with Pompe disease who are followed at Ruth Children's Hospital will be evaluated. Diagnosis is confirmed in all cases by deficient GAA activity in cultured fibroblasts or by Ultra Performance Liquid Chromatography - Tandem Mass Spectrometer (UPLC-MS/MS) in DBS and mutational analysis of genomic DNA, isolated from peripheral blood leukocyte.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2018-06-24 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 1-6 years
  Oxygen uptake evaluated by cardiopulmonary exercise testing (CPET)

SECONDARY OUTCOMES:
Six minute walk test | 1-6 years
  The distance gained after six minute of habitual walking.
Motor function test | 1-6 years
  Motor function test (GMFM-88) as assessed by experience physiotherapy.
GAA enzyme level | 1-6 years
  Self-collected blood samples (on a Guthrie card) for lysosomal enzyme acid alpha-glucosidase (GAA) blood levels.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Principal Investigator — Rambam
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
IPD is not planned to be available.